CLINICAL TRIAL: NCT06686667
Title: The Effect of Overnight Time Restricted Eating on Glucose Regulation in Rotating Shift Workers - A Randomised Controlled Feasibility Trial
Brief Title: The Feasibility of Overnight Time Restricted Eating and Impact on Glucose Levels in Shift Workers
Acronym: TREsh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: South Eastern Sydney Local Health District (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/ETH01526
Record Dates: First submitted 2024-11-04; First posted 2024-11-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Shift Work; Eating Behaviors
Keywords: Shift Worker Health; dietary intervention; time restricted eating; feasibility
MeSH Terms: conditions — Feeding Behavior; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Open label trial assessing a behavioral eating intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (Experimental): Participants will follow a time-restricted eating diet during day and night shifts over 2 weeks
  Interventions: Behavioral: Time Restricted Eating
- Control Arm (No Intervention): Participants will follow their usual eating patterns without restrictions during day and night shifts over 2 weeks

INTERVENTIONS:
Behavioral: Time Restricted Eating — The intervention arm will consist of a time-restricted eating protocol with fasting between 11:00 PM to 6:00 AM. Ad libitum eating will be allowed outside these times and the protocol will be administered during day and night shifts over a 2 week period.
  Arms: Time Restricted Eating

SUMMARY:
The aim of this clinical trial is to assess whether it is feasible for shift workers to follow a time-restricted eating diet. The trial will investigate the impact of time-restricted eating on blood glucose levels during day and night shifts both with and without the time-restricted eating diet.

The trial aims are:

* Is it feasible for shift workers to adhere to a night time time-restricted eating protocol?
* How does time-restricted eating affect blood glucose levels during the day and night shifts and over the whole day?

DETAILED DESCRIPTION:
Shift work is an essential component of modern workforces, with about 20% of the workforce regularly engaged in shift work. Research has shown shift workers are at higher risk of chronic diseases, including cardiometabolic disease, compared to day-only workers. Specifically, evidence shows eating overnight significantly increases the risk of metabolic syndrome. We also know eating patterns of shift workers and non-shift workers are different with evidence from our research showing shift workers engaged in night shift change their eating behaviors compared to day shifts. With a substantial proportion of the workforce involved in shift work, understanding the health challenges is crucial for developing targeted interventions and promoting a healthier shift working population.

Despite the need for behavioural eating interventions in shift workers, there is a lack of studies examining how these eating interventions would be implemented in real world contexts. Some dietary interventions related to quantity, quality and timing of food in shift workers have been reported, including limiting the quantity of food with various macronutrient restriction and low-calorie meal replacements, improving the quality of food with dietary advice/counselling, and promoting healthier food choices with variable results.

With recent recognition of the timing of food consumption being an important factor of metabolic regulation, time restricted eating (TRE) offers a viable strategy for improving metabolic health. TRE is a chrono-nutritional strategy involving close alignment of meal timing with typical circadian physiology over 24-hour periods. Typically, this involves an eating window of approximately 8 hours, with no eating during the night. Evidence shows TRE improves alignment of the fasting/eating cycle with the central circadian pacemaker and initiating nutrient-sensing pathways to ensure nutrient homeostasis. Research has shown TRE is an effective chrono-nutritional intervention for weight reduction, improvements in HbA1c and insulin levels, reduced insulin resistance or enhanced insulin sensitivity, improved glucose tolerance and reduced mean fasting glucose and improved quality of life. However, using TRE has not been examined extensively in shift workers in real world settings.

A recent narrative review found only three studies had investigated TRE as a diet strategy for shift workers under real-life conditions and these studies were conducted in populations with limited exposure to shift work situations (e.g. rotating shift work). Therefore, research is required that investigates the feasibility of TRE during night shifts in rotating shift workers.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals engaged in rotating shift work, including night shifts;
* Aged 23-60 years;
* At least 12 months experience in shift work;
* Willing to wear continuous glucose monitor sensors;
* Willing to engage in time restricted eating.

Exclusion Criteria:

* Diagnosis of diabetes (Type 1 or 2), any bariatric surgery, coeliac disease, inflammatory bowel disease, endocrine disorders affecting glucose metabolism, current or history of eating disorder, any liver, kidney, or coronary heart disease, obese (BMI>35) or underweight (BMI< 18) or any severe or unstable chronic medical conditions or cancers;
* Currently taking medications known to interact with glucose metabolism, i.e. thyroxin, insulin sensitizers, glucocorticoids, or anti-depressants, weight loss medication;
* Undertaking current structured or restrictive dietary plan;
* Shift workers who routinely do not eat between 23:00 and 06:00 hours during night shift;
* Current or planned pregnancy or currently breast feeding;
* Consume three or more standard alcohol containing beverages on a single occasion almost every day;
* People who identify as having significant caffeine dependency and are unwilling to limit intake of calorie free energy drinks;
* People with planned travel over time zones during the study period
* Any contraindication to use of Abott FreeStyle Libre Pro glucose sensor (eg prescription of vitamin C, Salicylic acid or paracetamol - to be reviewed by study clinician).

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of time-restricted eating (TRE) among shift workers (Recruitment and Participation Rate) | From enrolment to end of treatment at 2 weeks
  Feasibility will be assessed through a composite of the following metrics:
  Recruitment and participation rate (%) will be assessed as the percentage of participants randomized from the screened population.
  Each component will be assessed separately but reported as contributing factors to the overall feasibility.
Feasibility of time-restricted eating (TRE) among shift workers (Adherence Rate) | Two weeks
  Feasibility will be assessed through a composite of the following metrics:
  Adherence rate (%) percentage of participants who comply with the TRE protocol over a 2-week period, determined using self-reports Each component will be assessed separately but reported as contributing factors to the overall feasibility.
Feasibility of time-restricted eating (TRE) among shift workers (Study Completion Rate) | Two weeks
  Feasibility will be assessed through a composite of the following metrics:
  Study completion rate (%) percentage of participants who complete the 2-week study period without dropping out.
  Each component will be assessed separately but reported as contributing factors to the overall feasibility.

SECONDARY OUTCOMES:
Blood glucose levels during the 2-week study period | 2 weeks
  * Average 24-hour glucose levels;
  * Nocturnal glucose levels;
  * Sleep time glucose levels;
  * Day and night shift levels.
Facilitators and barriers associated with adherence to time restricted eating | 2 weeks
  Only in the intervention arm, participants will be asked questions about issues about eating patterns during the time restricted eating including barriers and facilitators for maintaining the fasting period.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Gordon, PhD, Principal Investigator — Woolcock Institute of Medical Research and Macquarie University
Locations (1):
- The Sutherland Hospital, Caringbah, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
All data will be dei-dentified using a unique study ID.